CLINICAL TRIAL: NCT05740722
Title: Nicotinamide Riboside Supplementation In Progressive Multiple Sclerosis: A Randomised Controlled Trial: The NORSEMAN Study
Brief Title: Nicotinamide Riboside Supplementation In Progressive Multiple Sclerosis
Acronym: Norseman
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 492199
Record Dates: First submitted 2023-01-30; First posted 2023-02-23 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis; Progressive Multiple Sclerosis
Keywords: nicotinamid riboside
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: A randomised placebo-controlled trial. Experimental: Placebo Placebo vs study drug (Nicotinamid riboside 500 mg x 2 po)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): Placebo vs study drug
  Interventions: Dietary Supplement: Placebo
- Nicotinamid Riboside (Experimental): Placebo vs study drug
  Interventions: Dietary Supplement: Nicotinamid riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamid riboside — 500 mg x 2 po
  Arms: Nicotinamid Riboside
Dietary Supplement: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Nicotinamide riboside (NR) for treatment of patients with progressive multiple sclerosis.

The main question it aims to answer is:

• Does NR delay disability progression in progressive multiple sclerosis?

Participants will be treated with NR or placebo for 30 months,

DETAILED DESCRIPTION:
After being informed about the study and risks, all patients giving written informed consent will undergo a screening period to determine eligibility for study entry.

At baseline patients who meet the eligibility requirements will be randomised in a double- blinded manner (patient and investigator) in a 1:1 ratio to nicotinamide riboside (1000 mg daily) or placebo (once a day)

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of progressive MS (secondary; SPMS or primary; PPMS) according to the 2013 revisions of clinical course of multiple sclerosis and the 2017 revisions of the McDonald criteria.
* Aged 18-65 years.
* EDSS 3-6.5
* Able to perform T25FW test
* The participant must have documented evidence of disability progression observed during the 24 months before screening.
* With or without a stable disease modifying therapy during the last three months.
* Written informed consent for study participation.

Exclusion Criteria:

* A diagnosis of relapsing MS according to the revisions of the McDonald criteria
* Neoplastic disease at baseline
* Previous history of malignant melanoma or breast cancer
* Stable phase of a progressive disease course
* Pregnancy or lactating female patients
* Dementia or other neurodegenerative disorder at baseline visit
* Comorbidity (psychiatric or somatic) that precludes study participation
* Use of high dose vitamin B3 supplementation within 30 days of enrolment
* Genetically confirmed mitochondrial disease or metabolic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with sustained disability progression over the treatment period | Baseline to month 30
  Defined as an increase in either expanded disability status scale (EDSS), timed 25 foot -walk test (T25W) or 9-hole-peg test.
  EDSS is measured in scores from 0 - 10. The higher the score the less ambulatory ability. Progression is defined as an increase of >/=1.0 point if baseline EDSS is </= 5.5 or an increase of >/=0.5 point if baseline EDSS is >/= 5.5. Progression in T25WT and 9HPT is defined as an increase of 20% from baseline measures in minutes/seconds.

SECONDARY OUTCOMES:
To determine the efficacy of NR compared with placebo, as reflected by EDSS | Baseline to month 30
  Proportion of patients with sustained disability progression over the treatment period
To determine the efficacy of NR compared with placebo, as reflected by 25-footwalk | Baseline to month 30
  Proportion of patients with sustained disability progression over the treatment period
To determine the efficacy of NR compared with placebo, as reflected by 9-Hole Peg test | Baseline to month 30
  Proportion of patients with sustained disability progression over the treatment period
To determine the efficacy of NR compared with placebo, as reflected by total volume of T2 lesions on MRI scans of the brain | Baseline to month 24
  MRI
To determine the efficacy of NR compared with placebo, as reflected by formation of lesions | Baseline to month 24
  MRI
Changes in brain atrophy in NR-treated patients with primary progressive multiple sclerosis as compared with placebo | Baseline to month 24
  MRI
Time to onset of sustained disability progression over the treatment period | Baseline to month 30
  Increase in either EDSS, T25FW or 9HPT that is sustained for at least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kjell-Morten Myhr, Study Director — Haukeland University Hopsital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No